CLINICAL TRIAL: NCT03384537
Title: Antimicrobial Effect of Tropolone Containing Versus Tropolone Free Mouthwash - Randomized Clinical Trail
Brief Title: Antimicrobial Effect of Tropolone Containing Versus Tropolone Free Mouthwash
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Awad Mohamed Abdelkadir, Master Degree, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-11-45
Record Dates: First submitted 2017-12-12; First posted 2017-12-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Dental Diseases
Keywords: intra-oral microorganisms.; cariogenic microorganisms
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: The participants in this study will be randomly divided into two groups according to the application of the mouth rinse agent (M); the first group M1) The participants will use Tropolone containing as a mouth rinse, the second group (M2) The participants will use chlorhexidine 0.2% as a mouth rinse.
  Then each participant will be monitoring at the base line T0: before using any mouthwash, T1: immedially after using tested mouthwash, T2: after one week and finally, T3: after two weeks of using the tested mouthwash.
  Each participant will be the reference/counted for self as a record.
Who Masked: Outcomes Assessor
Masking Description: A third party will perform the allocation sequence and assign the participants to rinsing agent in sequentially numbered opaque envelop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listerine total care zero (Experimental): Listerine total care zero
  Interventions: Combination Product: Listerine total care zero
- Chlorhexidine Mouthwash (0.2%). (Active Comparator): Chlorhexidine Mouthwash (0.2%).
  Interventions: Combination Product: Chlorhexidine Mouthwash (0.2%).

INTERVENTIONS:
Combination Product: Listerine total care zero — reducing intra-oral cariogenic microorganism.
  Arms: Listerine total care zero
Combination Product: Chlorhexidine Mouthwash (0.2%). — Chlorhexidine Mouthwash (0.2%).
  Arms: Chlorhexidine Mouthwash (0.2%).

SUMMARY:
The objective of this study is to compare the effect of Tropolone containing mouthwash versus CHX 0.2% mouthwash in reducing intraoral microorganism. Randomized clinical trial study

DETAILED DESCRIPTION:
Dental Caries disease prevented through the antibacterial mouthwash.

The prevalence of dental caries disease continues to be a challenge for oral health care professionals to this day.

In fact an alarming 92% of US adults (aged 20 to 64 years) have a history of dental caries. While strides have been made since the early 1970s the problem persists.

From the mid1990s until 2004 according to the National Health and Nutrition examination survey there was a small but significant increase in primary decay. This trend was even more severe in younger.

Dental Caries disease are not being treated can eventually turn into more serious issues. Fluoride has long been known as one of the key components to good oral health and the prevention of dental caries disease. It is a naturally occurring mineral that makes tooth enamel more resistant to acid producing bacteria that cause dental caries disease while also repairing teeth in the very early microscopic stages. While the use of fluoride in toothpaste has been responsible for a drop in dental caries disease since 1960 this significant problem still persists.

Yet, many people do not realize that also using a mouth rinse can result in 50% stronger teeth than brushing with fluoride toothpaste alone. The American Dental Association (ADA) recommends the use of mouth rinses with fluoride to help resist tooth decay. However, while it may appear so on the surface, not all fluoride mouth rinses are created the same.

At the Listerine brand, our commitment to innovation led to the creation of unique anti-cavity mouth rinses powered by breakthrough science called rapid fusion technology a unique fluoride delivery system which binds calcium ions with fluoride to create fluoride reservoirs that attach to tooth enamel and are then released over time for a greater fluoride uptake and greater enamel content of fluoride to the tooth surface.

Rapid fusion technology provides fluoride in a safe acidic environment that rapidly liberates calcium and phosphate ions. These ions combine to create millions of tiny fluoride reservoirs on tooth enamel and in saliva increasing the amount of fluoride on the tooth surface.

Throughout the day as enamel is exposed to acids from dietary sugars, the reservoirs dissolve and release fluoride to re-mineralize the teeth. The fluoride then binds to areas of weak demineralized enamel and attracts calcium and phosphate from saliva.

These ions penetrate the enamel and combine with fluoride to create a new stronger and more acid resistant mineral surface. In this way Rapid fusion technology enhances re-mineralization and inhibits demineralization of tooth enamel to provide. stronger teeth than brushing with fluoride toothpaste alone and greater re-mineralization of enamel.

The antimicrobial mouthwash is proved to prevent the development of dental plaque. The use of antimicrobial agents will lead to the avoidance of side effects complained by patients associated with the use of chlorhexidine.

And proving their potency against mutans streptococci will dramatically improve the oral health of patients as it is the major cause of dental plaque.

Dental plaque is reported to be a major health problem in public.

Therefore, reducing the incidence of caries disease through the use of antimicrobial agents will decrease the number of visits of patients complaining of plaque and associated health problems. Also, complaints of patients regarding side effects of will be of no concern to dentists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be between 18- 45 years of age.
2. All the volunteers participated in this study will be healthy looking with free medical history.
3. The volunteers will be asked to suspend their usual oral hygiene practice from two to four days before experiment studying.

Exclusion Criteria:

1. Patients with a compromised medical condition.
2. Volunteers that receive any antimicrobial agent during at least two weeks prior to study.
3. Volunteer with fixed, removable prosthesis or orthodontics appliance.
4. Volunteers with DMF above six will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial count. | Change from the baseline immediate after using mouthwash, at one week after mouthwash and at two weeks after regular use of mouthwash
  viability counts of Mutans Streptococci lactobacilli

CONTACTS AND LOCATIONS:
Overall Officials: Abdelkadir, Principal Investigator — Study Principal Investigator
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BACKGROUND:evaluate the antiplaque effects of an alcohol-free essential oil (alcohol-free EO) mouthwash and an amine fluoride/stannous fluoride with zinc lactate (SnFl-Zn) mouthwash compared to a positive control of chlorhexidine (CHX) mouthwash, using — https://www.ncbi.nlm.nih.gov/pubmed/?term=Efficacy+of+two+mouthwashes+on+3%E2%80%90day+supragingival+plaque+regrowth%3A+a+randomized+crossover+clinical+trial%E2%80%8F
- See also: Results:demonstrate that the phenols and their concentrations as contained within Listerine® could be further optimized in terms of selecting those which increase their general effectiveness, at concentrations that do not induce harm. — https://www.ncbi.nlm.nih.gov/pubmed/?term=A+preliminary+investigation+on+the+antimicrobial+activity+of+Listerine%C2%AE%2C+its+components%2C+and+of+mixtures+thereof%E2%80%8F

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03384537/Prot_SAP_001.pdf